CLINICAL TRIAL: NCT00776659
Title: An Observational Study Of Indian Breast Cancer Patients Receiving Adjuvant Therapy With Aromasin
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5991088
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-09

CONDITIONS: Breast Neoplasms
Keywords: An Observational Study of Indian Breast Cancer Patients Receiving Adjuvant Therapy with Aromasin; Antineoplastic Hormonal Drugs; Aromasin
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational
  Interventions: Other: Aromasin

INTERVENTIONS:
Other: Aromasin — Non-Interventional study design.
  Other Names: exemestane

SUMMARY:
To generate the following data from patients with early breast cancer treated with Aromasin® in the adjuvant setting in India.

* Efficacy of the treatment with Aromasin®
* Safety of the treatment with Aromasin®

DETAILED DESCRIPTION:
NA The study was prematurely discontinued due to slow enrollment and keeping in mind the observational nature of the study. The decision to terminate had been taken on 16th June 2012 and the LSLV occured on 14th September, 2012. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early breast cancer receiving adjuvant therapy with Aromasin® will be eligible.

Exclusion Criteria:

* Patients presenting with in situ cancers, recurrent or metastatic breast cancer, or a 2nd primary will not be included.
* Patients with a known hypersensitivity to Exemestane or its metabolites will also not be included.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early breast cancer receiving adjuvant therapy with Aromasin® will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- India (3):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Lucknow, Uttar Pradesh

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5991088&StudyName=An%20Observational%20Study%20Of%20Indian%20Breast%20Cancer%20Patients%20Receiving%0AAdjuvant%20Therapy%20With%20Aromasin%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- Exemestane: Exemestane (Aromasin) in accordance with local product document (LPD) and dose was adjusted according to medical and therapeutic necessity up to 3.5 years of duration or until tumor relapse occurred.
Period: Overall Study
Arm/Group | Exemestane
Started | 39
Completed | 13
Not Completed | 26
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 10
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Exemestane
Number analyzed (Participants) | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Locoregional/Distant Recurrence of Primary Breast Cancer
Description: Locoregional recurrence was defined as any recurrence of the breast cancer in the ipsilateral breast, chest wall or axillary lymph nodes.
Time Frame: Baseline until locoregional/distant recurrence of primary breast cancer (up to Year 3.5)
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of aromasin therapy. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 7
participants
  Locoregional/Distant Recurrence | 0
  Missing/No response | 1

2. Primary Outcome: Number of Participants With Appearance of Second Primary or Contralateral Breast Cancer
Time Frame: Baseline until appearance of second primary or contralateral breast cancer (up to Year 3.5)
Population: FAS included all enrolled participants who received at least 1 dose of aromasin therapy. 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 7
participants
  Second primary or contralateral breast cancer | 0
  Missing/No response | 1

3. Primary Outcome: Number of Participants Who Died
Time Frame: Baseline until death (up to Year 3.5)
Population: FAS included all enrolled participants who received at least 1 dose of aromasin therapy.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 39
participants | 0

4. Primary Outcome: Number of Participants Who Discontinued Aromasin Therapy
Time Frame: Baseline until discontinuation (up to Year 3.5)
Population: FAS included all enrolled participants who received at least 1 dose of aromasin therapy.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 39
participants | 26

5. Primary Outcome: Number of Participants With Gynecological, Cardiac, Thromboembolic, Musculoskeletal and Menopausal Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Number of participants with AEs related to gynecological, cardiac, venous thromboembolic, musculoskeletal and menopausal symptoms were reported. Gynecological AEs: bleeding, discharge, uterine dilatation and curettage; cardiac AEs: myocardial infarction, hypertension; musculoskeletal: joint stiffness, arthralgia, muscle cramps, fractures; menopausal symptoms: hot flushes, anxiety, depression, headache.
Time Frame: Baseline up to 28 days after last dose of study treatment
Population: FAS included all enrolled participants who received at least 1 dose of aromasin therapy.
Measure: Number; unit: participants
Arm/Group | Exemestane
Number analyzed (Participants) | 39
participants
  Gynecological AEs | 0
  Cardiac AEs | 0
  Venous thromboembolic events | 0
  Musculoskeletal AEs | 0
  Menopausal symptoms | 2

6. Primary Outcome: Change From Baseline in High Density Lipoprotein-Cholesterol (HDL-C), Low Density Lipoprotein-Cholesterol (LDL-C), Total Cholesterol and Triglycerides at Month 6, 12, 18, 24, 30, 36 and 42
Time Frame: Baseline, Month 6, 12, 18, 24, 30, 36, 42
Population: Results for this outcome were not reported because change from baseline in HDL-C, LDL-C, total cholesterol and triglycerides could not be calculated as no participant had data available at more than 1 time point.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

7. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) at Month 6, 12, 18, 24, 30, 36 and 42
Time Frame: Baseline, Month 6, 12, 18, 24, 30, 36, 42
Population: Results for this outcome were not reported because change from baseline in BMD could not be calculated as no participant had data available at more than 1 time point.
Arm/Group | Exemestane
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Exemestane
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 10/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane (N=39)
Abdominal distension (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 2
Lymphoedema (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Study was terminated due to slow enrollment and observational nature of the study. Low number of participants enrolled was not sufficient to conduct the planned analysis. Study was not terminated due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.